CLINICAL TRIAL: NCT00409214
Title: A Phase IIa Safety and Light Dose-escalation Study in Patients With Primary or Recurrent/High-grade Glioma (Defined for the Purposes of the Protocol as Anaplastic Astrocytoma [AA] or Glioblastoma Multiforme [GBM]) Using the Litx™ System to Confirm the Zone of Tumor Destruction During the Intraoperative Treatment of Glioma
Brief Title: Phase IIa Safety and Light Dose-escalation Study in Patients With Primary or Recurrent/High-grade Glioma Using the Litx™ System to Confirm the Zone of Tumor Destruction During the Intraoperative Treatment of Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSO-OL007
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: Glioma; Litx™; LS11; Glioblastoma multiforme; Anaplastic Astrocytoma; GBM; AA
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — Talaporfin

INTERVENTIONS:
Drug: LS11 (talaporfin sodium)
Device: Light source (interstitial light emitting diodes)
Procedure: Intraoperative placement of device in glioma

SUMMARY:
The pupose of this study is to demonstrate the safety of the Litx™ therapy and confirm the zone of tumor destruction with escalated light doses following intraoperative treatment of primary or recurrent glioma.

DETAILED DESCRIPTION:
Light Infusion Technology (Litx™) is a locoregional cancer treatment in which a systemically administered light-activated drug (LS11) is activated locally by illuminating the diseased tissue using light-emitting diodes (LEDs) of a specific wavelength. The activated photosensitizer reacts with endogenous oxygen to yield highly reactive species of oxygen that cause destruction of cellular structures such as mitochondria, lysosomes and cell walls leading to irreversible cell damage and tissue death.

Either twenty-four or twelve hours prior to surgery, the patient will receive an intravenous dose of 1 mg/kg of LS11, given IV by slow push over 3-5 minutes.

Following craniotomy, patients will undergo intraoperative placement of a single Light Source, centrally placed within the tumor, under direct visualization prior to tumor resection. Following placement of the light source (with the depth of the end of the light bar from the cortical surface to be calculated from the pre-operative MRI and spiral CT scan, so as to be centralized within the main tumor bulk), light will be delivered following a predetermined escalation schedule (either 100 J/cm or 200 J/cm) at 20 mW/cm light energy for a treatment time of 1 hour 24 minutes (100J/cm) or 2 hours 46 minutes (200 J/cm). The Light Source will then be manually removed and the tumor maximally resected.

The resected tumor and marginal tissue will be submitted for pathology to determine depth of cell death, extent of tumor tissue containing closed vessels, any evidence of vessel closure or other damage to tissues outside of the projected kill zone.

ELIGIBILITY:
Inclusion Criteria:

* Have primary or recurrent glioblastoma multiforme (GBM) or anaplastic astrocytoma (AA) undergoing planned tumor resection
* Have a right sided, supratentorial frontal or temporal lobe tumor
* Have right hand dominance
* Be adults aged >18 years
* Have a Karnofsky Performance Status score >70
* Have a estimated life expectancy of >12 weeks
* Have completed any prior antineoplastic therapy at least 4 weeks prior to surgery and be recovered from acute side effects
* Must have the understanding and ability to sign an informed consent document
* Be male or non-pregnant, non-lactating females. Patients who are fertile must agree to use an effective method of contraception during participation in the study
* Have a negative serum or urine pregnancy test within 14 days prior to treatment (if patient is a female of childbearing potential).

Exclusion Criteria:

Patients must be excluded if any of the following apply:

* Have tumors <2 cm in diameter
* Have inadequate organ function as evidenced by: PT or PTT >1.5 × control ; Platelet count <100,000/mm3 ; WBC <2,500/mm3 ; Neutrophils <2000/mm3 ; Hemoglobin <9 g/dL
* Be concurrently participating in another clinical trial involving experimental treatment
* Have any concurrent diseases or conditions that in the opinion of the investigator impair the patient's ability to complete the trial such as psychological, familial, sociological, geographical or medical conditions which in the Principal Investigator's opinion could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial's data are excluded.
* Have psychological, familial, sociological, geographical, or medical conditions which, in the Investigator's opinion, could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial data.
* Have a known sensitivity to porphyrin-type drugs or known history of porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety of the Litx™ therapy and confirm the zone of tumor destruction with escalated light doses following intraoperative treatment of primary or recurrent glioma

CONTACTS AND LOCATIONS:
Overall Officials: Sy-Shi Wang, PhD, Study Director — Light Sciences Oncology
Locations (1):
- Institute of Neurosurgery, Clinical Centre Serbia, Belgrade, Serbia